CLINICAL TRIAL: NCT06661733
Title: A Phase I Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Assess the Pharmacokinetics, Safety and Tolerability of AZD5462 in Participants With Renal Impairment
Brief Title: A Study to Investigate the Pharmacokinetics, Safety and Tolerability of AZD5462 in Participants With Renal Impairment
Acronym: GLITTER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9090C00010; 2024-514359-14-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Renal Impairment
Keywords: Renal impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with severe renal impairment (eGFR ≥ 15 to < 30 mL/min/1.73 m2, not requiring dialysis).
  Interventions: Drug: AZD5462
- Cohort 2 (Experimental): Participants who are healthy control (eGFR ≥ 90 mL/min/1.73 m2) matched at a group level to Cohort 1.
  Interventions: Drug: AZD5462
- Cohort 3 (conditional) (Experimental): Participants with moderate renal impairment (eGFR ≥ 30 to < 60 mL/min/1.73 m2).
  Interventions: Drug: AZD5462

INTERVENTIONS:
Drug: AZD5462 — Participants will receive AZD5462 orally.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), safety, and tolerability of AZD5462 in participants with impaired renal function.

DETAILED DESCRIPTION:
This is a Phase I, single dose, non-randomised, open-label, parallel group study to assess the PK, safety, and tolerability of AZD5462 in male and female participants (females of non-childbearing potential) with renal impairment.

This study consists of 3 cohorts:

1. Cohort 1: Participants with severe renal impairment (eGFR ≥ 15 to < 30mL/min/1.73 m2, not requiring dialysis).
2. Cohort 2: Participants who are healthy control (eGFR ≥ 90 mL/min/1.73 m2) matched at a group level to Cohort 1.
3. Cohort 3 (conditional): Participants with moderate renal impairment (eGFR ≥ 30 to < 60mL/min/1.73 m2).

This study comprises of three periods:

* Screening period: 21 days
* In-patient (Treatment) period: 4 days
* Out-patient visit: On Day 4, participants will return to the study site to undergo safety assessments and provide blood samples 72 hours post-dose. Participants may stay at the study site for this visit if preferred.
* Follow-up visit: On Day 7 (± 2), participants will return to the study site for safety assessments.

The duration of the study for an individual participant from the Screening Visit to the Follow-up Visit will be approximately 4 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

Healthy matched participants (cohort2):

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Stable renal function (eg, no clinically significant change in an eGFR within 3 months or longer prior to study screening), as determined by the investigator.
* An eGFR of ≥ 90 mL/min/1.73 m2, as determined at Screening Visit using the CKD-EPI 2021 creatinine only equation.

Participants With Renal Impairment:

* Participants with severe renal impairment (Cohort 1) must have an eGFR ≥ 15 to < 30 mL/min/1.73 m2, as determined at Screening Visit using the CKD-EPI 2021 creatinine only equation and not on dialysis.
* Participants with moderate renal impairment (Cohort 3) must have an eGFR of ≥ 30 to < 60 mL/min/1.73 m2, as determined at Screening Visit using the CKD-EPI 2021 creatinine only equation and not on dialysis.
* Stable renal impairment (eg, no clinically significant change in eGFR within 3 months or longer prior to study screening), for both Cohorts 1 and 3, as determined by the investigator.
* BMI within the range ≥ 18 to < 35 kg/m2, inclusive.
* Females of non-childbearing potential and males.

Main Exclusion Criteria:

* As judged by the investigator, any evidence of clinically significant disease or abnormal findings in screening assessments which in the investigator's opinion makes it undesirable for the participant to participate in the study.
* Positive HCV Ab, HBsAg, or HBcAb, HIV at screening.

Healthy Matched Participants (Cohort 2):

• Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment, or coagulation disorders) which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the result of the study, or the participant's ability to participate in the study.

Participants With Renal Impairment:

* Presence of unstable medical (eg, diabetes) or psychological conditions which, in the opinion of the investigator, would compromise the participant's safety or successful participation in this study.
* Renal transplant participants, participants on dialysis, and those with a history of acute kidney injury. Use of concurrent medication, which affects creatinine clearance such as cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine, quinine within 7 days of Day -1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | Day 1 to Day 4
  The AUCinf of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 to Day 4
  The AUClast of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Time to reach maximum observed plasma concentration (tmax) | Day 1 to Day 4
  The tmax of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Maximum observed plasma concentration (Cmax) | Day 1 to Day 4
  The Cmax of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Terminal elimination rate constant (λz) | Day 1 to Day 4
  The λz of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Terminal elimination half-life (t½λz) | Day 1 to Day 4
  The t½λz of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Apparent total body clearance (CL/F) | Day 1 to Day 4
  The CL/F of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Non-renal clearance of drug from plasma (CLNR/F) | Day 1 to Day 4
  The CLNR/F of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 to Day 4
  The Vz/F of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.
Renal clearance of drug (CLR) | Day 1 to Day 2
  The CLR of a single oral dose of AZD5462 in participants with renal impairment compared with healthy control participants matched at a group level will be assessed.

SECONDARY OUTCOMES:
Number of participants with Adverse Event (AEs) | Day 1 to Day 7
  The safety and tolerability of a single oral dose of AZD5462 in participants with renal impairment and healthy control participants matched at a group level will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes",indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9090C00010&attachmentIdentifier=bbe72919-8d24-4f84-bc0e-7174536e3742&fileName=d9090c00010__Redacted_CSR_synopsis.pdf&versionIdentifier=
- See also: results posted on www.astrazenecaclinicaltrials.com — https://www.astrazenecaclinicaltrials.com/study/D9090C00010/